CLINICAL TRIAL: NCT02534389
Title: Fish Oil Supplement Combined With Neoadjuvant Chemoradiation for Locally Advanced Rectal Cancer
Brief Title: Fish Oil Supplement in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1818/2013
Record Dates: First submitted 2015-08-17; First posted 2015-08-27 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; inflammation; omega-3; fish oil; nutritional status
MeSH Terms: conditions — Rectal Neoplasms; Inflammation | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fish oil group (Experimental): 4 soft gel with omega-3 fish oil
  Interventions: Dietary Supplement: omega-3 fish oil
- control group (No Intervention): without intervention

INTERVENTIONS:
Dietary Supplement: omega-3 fish oil — 2,4g of EPA + DHA
  Arms: fish oil group

SUMMARY:
Neoadjuvant treatment with radiotherapy (RDT) and chemotherapy (CT) are the treatment of choice for rectal adenocarcinomas in stages II and III. This results currently in pathologic complete response in 10% to 30% of cases. The immune and inflammatory response is altered in these individuals and is directly related to response to therapy. Both the disease and the treatment of colorectal cancer have an impact on quality of life and nutritional status. In studies with cells and animal models the incorporation of fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic (DHA) - derived from fish oil - has been shown to interfere in the process of inflammation, cell signaling and gene transcription enhancing the response to treatment. Are reported ability to restore the apoptosis of tumor cells, sensitization of tumor cells to chemotherapy, production of less pro-inflammatory cytokines and the preservation of normal energy and protein metabolism. The aim of this study is to verify if the daily consumption of 2.4 g EPA + DHA for adults in neoadjuvant therapy can promote changes on inflammatory and immunological markers of host response to tumor and if this response is altered by nutritional status. It is expected that supplementation can reflect in control of inflammatory and immune response in favor of tumor cell death contributes to pathological complete response and that it happens with preservation of nutritional status. Subjects will be randomized as to supplementation. All will be assessed in four moments during neoadjuvant therapy and immediate postoperative. Results will be presented by comparing the intervention group and control group at each moment.

ELIGIBILITY:
Inclusion Criteria:

* Candidate to neoadjuvant therapy according AC Camargo Cancer Center protocol;
* Accept consume fish oil capsules and participate in clinical, pathological and nutritional assessments by signing the consent form.

Exclusion Criteria:

* Be allergic to fish and fish products,
* It has previously undergone treatment for colorectal cancer or in presence of other concomitant cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Check effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on Glasgow Prognostic Score (GPS). | 18 months
  Combination of C-reactive protein and albumin, the Glasgow Prognostic Score (GPS), had independent prognostic value in patients with cancer. The GPS is the most extensively validated of the systemic inflammation-based prognostic scores and may be used in the routine clinical assessment of patients with cancer.

SECONDARY OUTCOMES:
Check effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on body weight and body composition with regard to skeletal muscle mass, and adipose tissue. | 18 months
  Measures: weight (kg) / Muscle mass (Kg) / adipose mass (Kg). Involuntary weight loss is common among patients with advanced cancer, contributing to poor treatment response, functional decline, and decreased survival. Nutritional intervention with fish oil may prevent deterioration of body composition.
Check for effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on muscle function. | 18 months
  Measure: hand grip strength (kg). Muscle function, assessed by hand grip strength, has been reported to be closely related to body composition and even more to muscle mass loss (sarcopenia).
Check for effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on quality of life (QOL). | 24 months
  Measured: specific oncologic questionnaire (EORTC QLQ-C30). The amount of symptoms distressed experienced by an individual has been related to QoL in a number of people with cancer. QoL is increasingly being used as a primary outcome measure in studies to evaluate the effectiveness of treatment.
Check for effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on inflammatory cytokines (IL-6, IL-1, TNF-alpha). | 18 months
  Measures: IL-6/ IL-1 / TNF-alpha. The cytokines interleukin-6 (IL-6), tumor necrosis factor alpha (TNFalpha) and interleukin-1 beta (IL-1beta) are critical mediators of the inflammatory response. Evidence has linked elevated levels of inflammatory cytokines with both loss of weight and therapeutical response.
Check for effects of daily consumption of 2.4 g of EPA + DHA for adults with rectal adenocarcinoma in neoadjuvant chemoradiation treatment on pathological response. | 24 months
  measure: pathological response grade. Pathological complete response after neoadjuvant chemoradiation and radical surgery in patients with locally advanced rectal cancer predicts better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Aguiar Jr., PhD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil